CLINICAL TRIAL: NCT01194830
Title: A Phase IIIb, 24-week, Randomised, Placebo-controlled, Double-blinded, Efficacy and Safety Study of Linagliptin (BI 1356) in Black/African American Patients With Type 2 Diabetes With a MTT Sub-study
Brief Title: Efficacy and Safety of Linagliptin (BI 1356) in Black/African Americans With Type 2 Diabetes With a MTT Sub-study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.75
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- Linagliptin (Active Comparator): 1 Tablet PO QD
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): 1 Tablet PO QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linagliptin — Active drug 1 tablet PO QD
  Arms: Linagliptin
Drug: Placebo — 1 Tablet PO QD
  Arms: Placebo

SUMMARY:
Study of linagliptin vs. placebo in Black/African American patients with T2DM with a MTT sub-study

ELIGIBILITY:
Inclusion criteria:

1. Dated written informed consent that is in accordance with GCP and local legislation.
2. Male and female Black / African American patients
3. Diagnosis of type 2 diabetes at least 3 months prior to the informed consent.
4. HbA1c more than or equal to 7.5% and less than or equal to 11% at Visit 1.
5. Patients are currently treatment-naive or being treated with up to one oral antidiabetic medication. Antidiabetic medication is to be unchanged for at least 10 weeks prior to the informed consent.
6. Age more than 18 and less than 80 years at Visit 1 (Screening).
7. BMI (Body Mass Index) less than 45 kg/m2 at Visit 1.

Exclusion criteria:

1. Myocardial infarction (MI), stroke or transient ischemic attack (TIA) within 3 months of informed consent.
2. Type 1 diabetes.
3. Impaired hepatic function, defined by serum levels of either alanine aminotransferase (ALT, SGPT), aspartate aminotransferase (AST, SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined at Visit 1.
4. Known prior hypersensitivity or allergy to the investigational product or its excipients.
5. Treatment with insulin within 3 months prior to informed consent.
6. Treatment with anti-obesity drugs (e.g., sibutramine, orlistat, rimonabant) within three months prior to informed consent or initiating therapy during the study.
7. Any prior use of dipeptidyl peptidase-4 (DPP-4) inhibitors.
8. Glucagon-like peptide-1 (GLP-1) agonists are excluded 3 months prior to informed consent.
9. History of alcohol or drug abuse within 3 months prior to informed consent that would interfere with trial participation as assessed by the Investigator.
10. Participation in another trial with an investigational drug within 3 months prior to informed consent or during the study.
11. Pre-menopausal women (last menstruation less than 1 year prior to informed consent) who:

    * are nursing or pregnant
    * are not surgically sterile
    * or are of child-bearing potential and are not practicing an acceptable method of birth control or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include transdermal patch, intrauterine devices/systems (IUDs / IUSs), oral, implantable or injectable contraceptives, and vasectomised partners. No exceptions will be made.

    Hormonal birth control should have been in use for at least three months prior to signing informed consent and continue at least until the next menstrual period after completing the study.
12. Current treatment with chronic use of systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent.
13. History of bariatric surgery.
14. Patients who have demonstrated an inability to be compliant (80-120%) with the dosing regimen during the placebo run-in period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (93):
- United States (93):
  - 1218.75.059 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1218.75.054 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1218.75.035 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1218.75.101 Boehringer Ingelheim Investigational Site, Toney, Alabama
  - 1218.75.066 Boehringer Ingelheim Investigational Site, Little Rock, Alaska
  - 1218.75.008 Boehringer Ingelheim Investigational Site, Pell City, Alaska
  - 1218.75.071 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1218.75.018 Boehringer Ingelheim Investigational Site, Chino, California
  - 1218.75.081 Boehringer Ingelheim Investigational Site, Garden Grove, California
  - 1218.75.109 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.75.040 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1218.75.047 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1218.75.106 Boehringer Ingelheim Investigational Site, Bartow, Florida
  - 1218.75.098 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 1218.75.036 Boehringer Ingelheim Investigational Site, Chiefland, Florida
  - 1218.75.105 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1218.75.083 Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - 1218.75.002 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1218.75.080 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1218.75.065 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 1218.75.007 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.75.029 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.75.045 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.75.084 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.75.017 Boehringer Ingelheim Investigational Site, Ocala, Florida
  - 1218.75.012 Boehringer Ingelheim Investigational Site, Pinellas Park, Florida
  - 1218.75.074 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1218.75.076 Boehringer Ingelheim Investigational Site, South Miami, Florida
  - 1218.75.003 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1218.75.039 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1218.75.075 Boehringer Ingelheim Investigational Site, Tallahassee, Florida
  - 1218.75.100 Boehringer Ingelheim Investigational Site, Tamarac, Florida
  - 1218.75.015 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1218.75.103 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 1218.75.049 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1218.75.067 Boehringer Ingelheim Investigational Site, Calhoun, Georgia
  - 1218.75.016 Boehringer Ingelheim Investigational Site, Dunwoody, Georgia
  - 1218.75.063 Boehringer Ingelheim Investigational Site, Lawrenceville, Georgia
  - 1218.75.056 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 1218.75.026 Boehringer Ingelheim Investigational Site, Rosswell, Georgia
  - 1218.75.079 Boehringer Ingelheim Investigational Site, Sandy Springs, Georgia
  - 1218.75.034 Boehringer Ingelheim Investigational Site, Snellville, Georgia
  - 1218.75.001 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.75.055 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.75.069 Boehringer Ingelheim Investigational Site, Owensboro, Kentucky
  - 1218.75.044 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1218.75.108 Boehringer Ingelheim Investigational Site, Essex, Maryland
  - 1218.75.086 Boehringer Ingelheim Investigational Site, Brockton, Massachusetts
  - 1218.75.087 Boehringer Ingelheim Investigational Site, Watertown, Massachusetts
  - 1218.75.051 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1218.75.088 Boehringer Ingelheim Investigational Site, Flint, Michigan
  - 1218.75.099 Boehringer Ingelheim Investigational Site, Biloxi, Mississippi
  - 1218.75.006 Boehringer Ingelheim Investigational Site, Atco, New Jersey
  - 1218.75.004 Boehringer Ingelheim Investigational Site, Camden, New Jersey
  - 1218.75.031 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1218.75.095 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1218.75.038 Boehringer Ingelheim Investigational Site, Asheboro, North Carolina
  - 1218.75.009 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1218.75.023 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1218.75.060 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1218.75.005 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 1218.75.107 Boehringer Ingelheim Investigational Site, High Point, North Carolina
  - 1218.75.020 Boehringer Ingelheim Investigational Site, Jacksonville, North Carolina
  - 1218.75.027 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1218.75.096 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1218.75.090 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1218.75.078 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1218.75.037 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1218.75.082 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1218.75.010 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1218.75.028 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1218.75.091 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 1218.75.072 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1218.75.068 Boehringer Ingelheim Investigational Site, Greenwood, South Carolina
  - 1218.75.097 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1218.75.024 Boehringer Ingelheim Investigational Site, Brentwood, Tennessee
  - 1218.75.025 Boehringer Ingelheim Investigational Site, Collierville, Tennessee
  - 1218.75.011 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 1218.75.042 Boehringer Ingelheim Investigational Site, Humboldt, Tennessee
  - 1218.75.030 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1218.75.050 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1218.75.053 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.75.057 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.75.064 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.75.104 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.75.043 Boehringer Ingelheim Investigational Site, Houton, Texas
  - 1218.75.022 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.75.058 Boehringer Ingelheim Investigational Site, Sugar Land, Texas
  - 1218.75.033 Boehringer Ingelheim Investigational Site, Tomball, Texas
  - 1218.75.102 Boehringer Ingelheim Investigational Site, Tomball, Texas
  - 1218.75.094 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 1218.75.092 Boehringer Ingelheim Investigational Site, Whitney, Texas
  - 1218.75.019 Boehringer Ingelheim Investigational Site, Virgnia Beach, Virginia

REFERENCES:
- [Derived] Lajara R, Aguilar R, Hehnke U, Woerle HJ, von Eynatten M. Efficacy and safety of linagliptin in subjects with long-standing type 2 diabetes mellitus (>10 years): evidence from pooled data of randomized, double-blind, placebo-controlled, phase III trials. Clin Ther. 2014 Nov 1;36(11):1595-605. doi: 10.1016/j.clinthera.2014.07.020. Epub 2014 Sep 16. PMID 25236917
- [Derived] Thrasher J, Daniels K, Patel S, Whetteckey J. Black/African American patients with type 2 diabetes mellitus: study design and baseline patient characteristics from a randomized clinical trial of linagliptin. Expert Opin Pharmacother. 2012 Dec;13(17):2443-52. doi: 10.1517/14656566.2012.740459. Epub 2012 Nov 8. PMID 23134211

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Tablet: Placebo matching linagliptin 5 mg tablet
- Linagliptin 5 mg Tablet: Linagliptin 5 mg (milligrams) tablet given by mouth once daily
Period: Overall Study
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Started | 124 | 110
Completed | 88 | 83
Not Completed | 36 | 27
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 5 | 4
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Non-compliance issues | 4 | 4
Not completed — Other Reason | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet | Total
Number analyzed (Participants) | 120 | 106 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] — 4 subjects in each treatment arm were excluded from analysis
  years | 54.1 (9.9) | 53.7 (10.1) | 53.9 (9.9)
Age, Customized [Number; unit: Number of participants] — 4 subjects in each treatment arm were excluded from analysis
  Number of participants
    < 65 years | 104 | 89 | 193
    65 to 74 years | 12 | 14 | 26
    >= 75 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants] — 4 subjects in each treatment arm were excluded from analysis
  Participants
    Female | 59 | 46 | 105
    Male | 61 | 60 | 121
Weight [Mean (Standard Deviation); unit: kilograms] — 4 subjects in each treatment arm were excluded from analysis
  kilograms | 99.02 (20.16) | 95.83 (20.96) | 97.52 (20.55)
Weight categories [Number; unit: Number of participants] — 4 subjects in each treatment arm were excluded from analysis
  Number of participants
    <= 70 kilograms | 2 | 8 | 10
    > 70 to 80 kilograms | 21 | 18 | 39
    > 80 to 90 kilograms | 25 | 26 | 51
    > 90 kilograms | 72 | 54 | 126
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter] — 4 subjects in each treatment arm were excluded from analysis
  kilograms per square meter | 33.35 (5.36) | 32.04 (6.10) | 32.74 (5.74)
Body Mass Index (BMI) categories [Number; unit: Number of participants] — 4 subjects in each treatment arm were excluded from analysis
  Number of participants
    < 30 kilograms/square meter | 33 | 45 | 78
    >= 30 kilograms/square meter | 87 | 61 | 148
Height [Mean (Standard Deviation); unit: centimeters] — 4 subjects in each treatment arm were excluded from analysis
  centimeters | 172.1 (10.9) | 172.8 (10.3) | 172.4 (10.6)
Waist circumference [Mean (Standard Deviation); unit: centimeters] — 4 subjects in each treatment arm were excluded from analysis
  centimeters | 111.5 (16.7) | 103.5 (20.2) | 107.7 (18.8)
Smoking status [Number; unit: Number of participants] — 4 subjects in each treatment arm were excluded from analysis
  Number of participants
    Never smoked | 82 | 56 | 138
    Ex-smoker | 22 | 21 | 43
    Currently smokes | 16 | 29 | 45
Alcohol status [Number; unit: Number of participants] — 4 subjects in each treatment arm were excluded from analysis
  Number of participants
    Non drinker | 70 | 61 | 131
    Drinks - no interference with study | 50 | 45 | 95
    Drinks - possible interference with study | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication and had both a baseline HbA1c value and an on-treatment HbA1c value. Four subjects in each arm excluded for site non-compliance.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 105 | 93
Percentage | -0.25 (0.16) | -0.84 (0.15)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0005, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and number of other Oral Antidiabetic Drugs; Least Squares Mean Difference = -0.58, 95% CI [-0.91 to -0.26], Standard Error of Mean 0.16

2. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 6 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 105 | 93
Percentage | -0.22 (0.10) | -0.64 (0.09)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and number of other Oral Antidiabetic Drugs; Least Squares Mean Difference = -0.42, 95% CI [-0.62 to -0.22], Standard Error of Mean 0.10

3. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 12 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 105 | 93
Percentage | -0.17 (0.14) | -0.72 (0.13)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0002, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and number of other Oral Antidiabetic Drugs; Least Squares Mean Difference = -0.55, 95% CI [-0.84 to -0.26], Standard Error of Mean 0.15

4. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 18 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 18 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 105 | 93
Percentage | -0.26 (0.14) | -0.81 (0.14)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0003, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and number of other Oral Antidiabetic Drugs; Least Squares Mean Difference = -0.55, 95% CI [-0.85 to -0.26], Standard Error of Mean 0.15

5. Secondary Outcome: Occurrence of Absolute Efficacy Response (HbA1c < 7%) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 110 | 98
Participants
  Responder (HbA1c < 7.0%) | 10 | 26
  Non-responder (HbA1c >= 7.0%) | 100 | 72
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 4.063, 95% CI 2-sided [1.764 to 9.358]

6. Secondary Outcome: Occurrence of Absolute Efficacy Response (HbA1c < 6.5%) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 110 | 98
Participants
  Responder (HbA1c < 6.5%) | 2 | 9
  Non-responder (HbA1c >= 6.5%) | 108 | 89
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0352, Regression, Logistic; Odds Ratio (OR) = 5.433, 95% CI 2-sided [1.124 to 26.260]

7. Secondary Outcome: Occurrence of Relative Efficacy Response (Reduction in HbA1c >= 0.5%) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 110 | 98
Participants
  Responder (reduction in HbA1c >= 0.5%) | 33 | 53
  Non-responder (reduction in HbA1c < 0.5%) | 77 | 45
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 2.951, 95% CI 2-sided [1.651 to 5.274]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 24 Weeks
Time Frame: baseline, 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication and had both a baseline FPG value and an on-treatment FPG value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL (milligrams per deciliter)
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 106 | 95
mg/dL (milligrams per deciliter) | -11.0 (6.6) | -22.9 (6.4)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0972, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c, baseline FPG, and number of other Oral Antidiabetic Drugs; Least Squares Mean Difference = -12.0, 95% CI [-26.1 to 2.2], Standard Error of Mean 7.2

9. Secondary Outcome: Change From Baseline in 2-hour Post-prandial Glucose (PPG) After 24 Weeks
Time Frame: baseline, 24 weeks
Population: Meal Tolerance Test, observed cases data set (MTT-OC) includes all randomized patients who participated in the MTT sub-study. Patients required to have both baseline and on-treatment results.
Measure: Least Squares Mean (Standard Error); unit: mg/dL (milligrams per deciliter)
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 11 | 10
mg/dL (milligrams per deciliter) | -36.77 (23.76) | -38.74 (22.77)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.9368, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c, baseline 2-hour PPG, and number of other Oral Antidiabetic Drugs; Least Squares Mean Difference = -1.97, 95% CI [-53.80 to 49.86], Standard Error of Mean 24.45

ADVERSE EVENTS:
Time Frame: 24 weeks (from day of first dose until 7 days after last dose)
Description: Four subjects in each treatment arm were excluded due to site non-compliance issues.
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Serious Adverse Events (participants affected / at risk) | 2/120 | 1/106
Other Adverse Events (participants affected / at risk) | 15/120 | 9/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tablet (N=120) | Linagliptin 5 mg Tablet (N=106)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tablet (N=120) | Linagliptin 5 mg Tablet (N=106)
Urinary tract infection (Infections and infestations) | 4 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 3

LIMITATIONS AND CAVEATS:
Eight randomized subjects were excluded from all analysis due to overall data integrity issues at the site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.